CLINICAL TRIAL: NCT07209930
Title: Inter- and Intraindividual Variability of the Acute Glucose Response to Exercise in Healthy Adults and People Living With Type 1 Diabetes: A Cross-over Replicate Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Collaborators: Taighde Éireann - Research Ireland (Unknown); Irish Research Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: LS-24-26-Merlo-Horner; EBPPG/2023/627 (Other Grant/Funding Number: Research Ireland)
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-08

CONDITIONS: Exercise; Healthy Participants; Glucose Variability; Type 1 Diabetes (T1D)
Keywords: reproducibility; exercise; Type 1 diabetes; glucose
MeSH Terms: conditions — Motor Activity; Diabetes Mellitus, Type 1 | interventions — Exercise; RE1-silencing transcription factor

STUDY DESIGN:
Intervention Model Description: Replicate crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise and Rest (Experimental): At the first test visit participants will complete 30 minutes exercise on a cycle ergometer, and at the second visit they will remain at rest. Identical conditions in an identical order will be repeated the following week.
  Interventions: Other: Exercise; Other: Rest
- Rest and Exercise (Experimental): At the first test visit participants will remain at rest and at the second visit they will complete 30 minutes exercise on a cycle ergometer. Identical conditions in an identical order will be repeated the following week.
  Interventions: Other: Exercise; Other: Rest

INTERVENTIONS:
Other: Exercise — After a 12h overnight fast, baseline measurements are collected. Participants are then provided with a standardized breakfast meal (60g carbohydrate). After consumption of the breakfast, participants remain seated seated for 30 minutes, before cycling on a cycle ergometer for 30 minutes at an intensity equivalent to 10% above the first ventilatory threshold (VT1). Sixty minutes of rest sitting on a chair will follow the 30-minute cycle.
  During the total 120 minute test, various measurements are collected at regular intervals, including: blood glucose measurements via finger prick, CGM measurements, RPE, HR, measures of heart rate variability (HRV) (RMSSD (Root Mean Square of Successive Differences) and SDNN (Standard Deviation of NN intervals)), and intensity of any hypoglycaemia-related symptoms using a Visual Analogue Scale (VAS).
Other: Rest — The procedure for the resting condition visits is identical to that of the exercise condition, with the only difference being that the 30-minute cycling session will be replaced by an additional 30 minutes of seated rest. This will ensure that the total duration of the session and the timing of all measurements will remain consistent across conditions.

SUMMARY:
The goal of this clinical trial is to investigate if blood glucose responses are similar between and within individuals in response to standardized exercise in adults with and without Type 1 diabetes. The main questions it aims to answer are:

What is the reproducibility of acute glycaemic responses to exercise within and between subjects in adults living with Type 1 Diabetes and in healthy adults? What is the agreement between glucose levels obtained by continuous glucose monitor (CGM) and blood glucose monitor?

Participants will cycle on a cycle ergometer or rest after consuming a standardized breakfast, while glucose levels are monitored by CGM and capillary blood sampling.

DETAILED DESCRIPTION:
This study follows a non-blinded randomized replicate crossover study design. The study involves two phases, one phase will involve participants with T1D and the other phase will involve healthy adults. The sample size will be approximately 12 in each phase. Both phases will follow the same protocol consisting of 2 arms (exercise (EX) and rest).

Participants will attend 5 visits in total in the laboratory. They will first undergo baseline assessments and maximal exercise testing before being randomized to receive either an exercise (EX) or resting (REST) condition at their visit first. The two visits will then repeated to assess reproducibility of the outcomes in the same order the following week (EX RE and REST RE). All test visits will be separated by a minimum washout period of 72 hours.

The first visit will last approximately 1 hour and involves signing informed consent, body composition assessment (BodPod), maximal exercise testing (Vo2 max) and completion of questionnaires.

Before each condition, participants are asked to refrain from strenuous physical activity and alcohol for at least 24 hours prior to the test(s). Prior to the first main testing day (either EX or RE based on randomization), participants are asked to record their dietary intake for 24h and asked to replicate it in the same period before the subsequent conditions.

Testing visits have a duration of 2 hours each. Participants will arrive at the laboratory after an overnight fast always at the same time in the morning (about 9am). While seated, baseline measurements will be collected, including 2 blood glucose measurements via finger prick, 2 CGM measurements, RPE, HR, measures of heart rate variability (HRV), and participants will the intensity of any hypoglycaemia-related symptoms using a Visual Analogue Scale (VAS). The same measurements will be repeated at regular intervals throughout the visit.

Participants were then provided with a standardized breakfast meal (60g of CHO) that they were instructed to consume within 10 minutes. After consumption of the breakfast, a clock was started. Participants remained seated for 30 minutes, and - during the EX condition - cycled on a cycle ergometer for 30 minutes at an intensity equivalent to 10% above VT. Sixty minutes of rest sitting on a chair follow the 30-minute cycle, before participants can leave the laboratory.

The procedure for the resting condition visits is identical to that of the exercise condition, with the only difference being that the 30-minute cycling session is replaced by an additional 30 minutes of seated rest. This ensures that the total duration of the session and the timing of all measurements remains consistent across conditions.

ELIGIBILITY:
Inclusion Criteria:

(Healthy and T1D phases):

* age between 18 and 60 years old;
* being healthy individuals;
* engagement in physical activity at least once a week; (T1D phase):
* diagnosis of T1D for >18 months;
* hypoglycaemia self awareness.

Exclusion Criteria:

(Healthy and T1D phases)

* presence of cardiovascular disease or contraindications to exercise;
* infectious or inflammatory conditions;
* chronic renal or liver disease;
* pregnancy;
* gestational diabetes;
* diagnosed eating disorders;
* any physical or mental condition preventing participation; (Healthy phase)
* diabetes mellitus (type 1 or type 2); (T1D phase)
* inability to self-manage diabetes.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Interstitial glucose | Over 2 hours: 2 samples at baseline in the fasted state before breakfast consumption; and every 5 minutes following breakfast for 2 hours.
  Interstitial glucose values (mmol/l) collected via Freestyle libre 2 Continuous Glucose Monitor
Capillary glucose | 2 hours: (1) at baseline before breakfast consumption; (2) every 10 minutes over 30 minutes after breakfast consumption during rest; (3) every 5 minutes for 30 minutes during cycle or seated rest based on intervention; (4) every 10 minutes for 60 min.
  Capillary glucose was measured via finger prick using a blood glucose monitor.

SECONDARY OUTCOMES:
Heart-rate variability | 2 hours: (1) at baseline before breakfast consumption. (2) every 10 minutes for 120 minutes. (3) extra measurements of HR only were taken during the second thirty minutes, resulting in HR measurements at 5-minutes intervals during that time-frame.
  Measures of heart rate variability including HR, RMSSD and SSND were collected using polar monitors and chest straps.
Perception of symptoms of Hypoglycaemia. | 2 hours: (1) at baseline before breakfast consumption; (2) every 20 minutes for 120 minutes.
  100 millimetre Visual Analogue Scales (VAS) will be used. This VAS has anchors located at each end of the scale. On the left end of the scale (0 mm), the "not at all" response is represented, while the right end (100 mm) represents the "extremely" response. Participants mark along the line where it most represents their subjective perception of 7 individual symptoms of hypoglycaemia (sweatiness; anxiety; hunger; thirst; difficulties in concentrating; blurred vision; dizziness) between both ends.
Reporting of Perceived Exortion (RPE) | 1 hour: (1) at baseline before breakfast consumption; (2) every 5 minutes during the second half hour.
  Ratings of Perceived Exertion (RPE) were collected using the Borg 6-20 Scale. Participants were initially familiarised with the scale during their baseline visit to ensure proper understanding.

CONTACTS AND LOCATIONS:
Locations (1):
- University College Dublin, Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
It is not approved within the ethics application to share IPD.